CLINICAL TRIAL: NCT01200030
Title: A Home-Based Program of Transcutaneous Electrical Nerve Stimulation and Task-Related Trunk Training Improves Trunk Control in Patients With Stroke: A Randomized Controlled Clinical Trial
Brief Title: Effects of Home-based Program in Improving Sitting Balance and Upper Limb Functions in Patients With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Shamay Ng, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DHSC_NG; DHSC_NG_001
Record Dates: First submitted 2010-09-10; First posted 2010-09-13 (Estimated); Results first posted 2019-01-04 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2018-07

CONDITIONS: Stroke
Keywords: Sitting balance; Stroke
MeSH Terms: conditions — Stroke | interventions — Electric Stimulation; Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- electrical stimulation with exercises (Experimental): The TENS + TRTT group received TENS simultaneously with the TRTT at home under the instruction of a physical therapist.
  Interventions: Behavioral: electrical stimulation with exercises
- placebo stimulation with exercises (Placebo Comparator): The TENS + TRTT group received placebo-simultaneously with the TRTT at home under the instruction of a physical therapist.
  Interventions: Behavioral: placebo stimulation with exercises
- Control (No Intervention): Subjects in this group did not receive any active training. Home safety advice and health education including diet control and blood pressure monitoring were given to the subjects during the home-visit and telephone follow-up.

INTERVENTIONS:
Behavioral: electrical stimulation with exercises — electrical stimulation with exercises
  Arms: electrical stimulation with exercises
Behavioral: placebo stimulation with exercises — placebo stimulation with exercises
  Arms: placebo stimulation with exercises

SUMMARY:
The investigators hypothesize that application of electrical stimulation would augment the effects of exercises in patients with stroke. Combined electrical stimulation with exercises for 6 weeks would lead to earlier and greater improvement in motor functions when compared with placebo-stimulation with exercises.

DETAILED DESCRIPTION:
Previous studies have shown that repeated sensory inputs from transcutaneous electrical stimulation (TES) could enhance brain plasticity and conical motor output. Home-based rehabilitation is shown to be effective in motor recovery and improvement of functional ability in stroke rehabilitation.

The aim of this study was to develop a home-based rehabilitation program to investigate whether combined electrically induced sensory inputs through TES with task-related trunk training (TRTT) in a home-based program would induce earlier and/or greater improvement in, seated reaching distance and trunk control when compared with placebo TES and TRTT, or control with no active treatment in subjects with chronic stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis with first stroke for more than 6 months
2. Discharge from all rehabilitation services
3. Ability to understand and follow commands
4. A carer able for helping the home program
5. No contraindication to assessment protocol and training

Exclusion Criteria:

1. Cognitive disorder with Abbreviated Mental Test less than 7
2. Unilateral neglect with Star cancellation Test less than 47
3. Sensory deficit
4. Unable to give informed consent
5. Unable to speak either Cantonese or English or Mandarin
6. Commodity that preclude them from undergoing training and assessment
7. Neurological disease other than stroke

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shamay Ng, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

RESULTS

PARTICIPANT FLOW:
Groups:
- Electrical Stimulation With Exercises: electrical stimulation with exercises: electrical stimulation with exercises (TES+ TRlT)
- Placebo Stimulation With Exercises: placebo stimulation with exercises: placebo stimulation with exercises (pTES+ TRlT)
- Control: No active treatment
Period: Overall Study
Arm/Group | Electrical Stimulation With Exercises | Placebo Stimulation With Exercises | Control
Started | 12 | 13 | 12
Completed | 12 | 13 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Electrical Stimulation With Exercises | Placebo Stimulation With Exercises | Control | Total
Number analyzed (Participants) | 12 | 13 | 12 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (10.7) | 56.3 (7.4) | 59.3 (10.4) | 57.8 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 3 | 10
  Male | 8 | 10 | 9 | 27
Region of Enrollment [Number; unit: participants]
  Hong Kong | 12 | 13 | 12 | 37

OUTCOME MEASURES:

1. Primary Outcome: Trunk Impairment Scale
Description: The Trunk impairment scale is a 2 to 4-point ordinal scale. The scale assesses static and dynamic sitting balance and trunk coordination. The maximum scores on the static sitting balance, dynamic sitting balance, and coordination subscales are 7, 10, and 6 points, respectively. The total score of Trunk impairment scale ranges between 0 and 23 points, with a higher score representing better trunk control. The static sitting balance subscale evaluated the trunk stability with both feet on the floor and with the legs crossed. The dynamic sitting balance subscale evaluated the ability to perform trunk side flexion. The coordination components evaluated the ability to selectively rotate the upper and lower parts of the trunk.
Time Frame: baseline, 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Electrical Stimulation With Exercises | Placebo Stimulation With Exercises | Control
Number analyzed (Participants) | 12 | 13 | 12
units on a scale
  Baseline | 13.2 (1.8) | 13.8 (1.3) | 13.9 (2.2)
  After training (6-week) | 19.0 (2.1) | 18.4 (1.5) | 15.2 (2.6)
Statistical Analysis 1: Comparison: Electrical Stimulation With Exercises vs Placebo Stimulation With Exercises vs Control; Null hypothesis: No significant differences existed between the percentage of change in Trunk Impairment Scale (TIS) score among the three groups; Test type: Other — The effect size of the intervention was adopted from a mate-analysis . The showed an average effect size of 0.59 in improving the motor control of limbs in people with stroke. A sample size for each group was set at 11 . Presuming that there would be a drop-out rate of 10% during the course of study, an extra 1 subject was recruited in each group. the sample size was 36. The statistical significance was set at 5% (alpha < 0.05) with power equal to 80%; p < 0.001, Kruskal-Wallis — Post-hoc pairwise comparisons have been conducted. Please refer to subsequent data analyses
Statistical Analysis 2: Comparison: Electrical Stimulation With Exercises vs Placebo Stimulation With Exercises; Post-Hoc pairwise comparison comparing the effects of electrical stimulation with exercises group and placebo stimulation with exercises group. Null hypothesis: There was no significant difference existed on the changes of the Trunk Impairment Scale score between the two groups; Test type: Other; p = 1.00, Wilcoxon (Mann-Whitney) — The p-value was adjusted for multiple comparisons. A p-value smaller than 0.05 indicated statistical significance
Statistical Analysis 3: Comparison: Electrical Stimulation With Exercises vs Control; Post-Hoc pairwise comparison comparing the effects of electrical stimulation with exercises group and control group. Null hypothesis: There was no significant difference existed on the changes of the Trunk Impairment Scale score between the two groups; Test type: Other; p = 0.002, Wilcoxon (Mann-Whitney) — The p-value was adjusted for multiple comparisons. A p-value smaller than 0.05 indicated statistical significance
Statistical Analysis 4: Comparison: Placebo Stimulation With Exercises vs Control; Post-Hoc pairwise comparison comparing the effects of placebo stimulation with exercises group and control group. Null hypothesis: There was no significant difference existed on the changes of the Trunk Impairment Scale score between the two groups; Test type: Other; p = 0.003, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Forward Sitting Functional Reach Test
Description: Sitting Functional Reach was used to assess the limits of stability in reaching activities. The sitting functional reach test measures how far forward, from a sitting position, a subject can bend forward to reach without losing his/her balance. A longer reaching distance indicated a better trunk control.
Time Frame: baseline, 6 weeks
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Electrical Stimulation With Exercises | Placebo Stimulation With Exercises | Control
Number analyzed (Participants) | 12 | 13 | 12
cm
  Baseline | 22.2 (6.9) | 28.7 (8.8) | 29.0 (9.5)
  After training (6 weeks) | 29.5 (5.2) | 34.1 (7.4) | 28.8 (7.2)
Statistical Analysis 1: Comparison: Electrical Stimulation With Exercises vs Placebo Stimulation With Exercises vs Control; Null hypothesis: No significant differences existed between the percentage of change in reaching distance between the three groups; Test type: Other; p = 0.055, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: from the start of training up to 4 weeks after training ended
Arm/Group | Electrical Stimulation With Exercises | Placebo Stimulation With Exercises | Control
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/13 | 0/12

LIMITATIONS AND CAVEATS:
The number of home-visit in transcutaneous electrical stimulation (TES)+ task-related trunk training (TRlT) group and placebo-TES (pTES) + TRlT group was greater than the control group who had no active treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No